CLINICAL TRIAL: NCT06074328
Title: Blended Reality Immersion for Geriatric Head Trauma: The BRIGHT Randomized Clinical Trial
Brief Title: Blended Reality Immersion for Geriatric Head Trauma: The BRIGHT Study
Acronym: BRIGHT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Mira Ghneim, Assistant Professor Program In Trauma, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HP-00105456
Record Dates: First submitted 2023-08-31; First posted 2023-10-10 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- No-VR Group (No Intervention)
- VR-Group (Experimental)
  Interventions: Device: Virtual Reality Neurocognitive Exercises administered through an Oculus Headset

INTERVENTIONS:
Device: Virtual Reality Neurocognitive Exercises administered through an Oculus Headset — Virtual Reality Neurocognitive Exercises administered through an Oculus Headset as a form of neurorehabilitation in patients who suffer a traumatic brain injury.
  Arms: VR-Group

SUMMARY:
Traumatic brain injury (TBI) is a major public health concern, particularly among older adults (OAs) ≥ 65 years of age. Each year in the United States, TBI results in over 600,000 emergency department visits and hospitalizations among OAs. Mild TBI (mTBI) accounts for 80% of all TBI in OAs and is quite understudied in this rapidly growing population. mTBI, is mild in name only, as it can result in dysfunction in multiple cognitive domains, including attention, processing speed, executive functioning and memory and has been shown to be associated with progressive brain atrophy and increased susceptibility to neurodegenerative disorders. Cognitive rehabilitation therapy is an evidence-based approach that can successfully improve cognitive impairment following TBI. Virtual reality (VR) is emerging as a technology that can assess cognitive impairment and provide a neurorehabilitation modality (NRM) to improve cognitive decline post TBI. Not only can VR provide a variety of environments like those encountered in real life and be adapted to varying levels and types of cognitive disability, but it can also be used safely in a patient's home with minimal equipment. Yet, despite the promise of cognitive rehabilitation using VR among OAs, very few studies to date have assessed the efficacy of VR cognitive rehabilitation in TBI. The aim of this study is to assess the effect and collect data on the efficacy and feasibility of a virtual reality application as a neurorehabilitation modality on executive functioning (attention, immediate memory, and visual-spatial skills) in OAs with mTBI. The hypothesis is that The use of VR mediated cognitive exercises post mTBI will be associated with improved executive function at 6-weeks post-randomization compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age or older
* Diagnosed with a mild traumatic brain injury
* Community dwelling
* English speaking
* Live within a 30 mile radius from the trauma center
* Active phone number
* Able to provide informed consent

Exclusion Criteria:

* Known history of cognitive impairment
* Known history of functional impairment
* History of seizure disorders
* Medical implantable devices ( pacemaker & defibrillator)
* Substance use disorder
* Other severe traumatic injuries to the neck, chest, abdomen, spine and pelvis

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-11-29 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Change in the immediate memory domain score on the Repeatable Battery for Neuropsychological Assessment | 7 weeks post enrollment
  individually administered test measuring attention, language, visuospatial/constructional abilities, and immediate and delayed memory. The SCORES range from 40-160 with a mean and standard deviation of 100 and 15. Higher score = better outcome

CONTACTS AND LOCATIONS:
Locations (1):
- R Adams Cowley Shock Trauma Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No